CLINICAL TRIAL: NCT06731426
Title: Effects of Multi-session, Personalized Cognitive Bias Modification for Thought-Action-Fusion Among Adults with Obsessive-Compulsive Symptoms: a Randomized Controlled Trial
Brief Title: Multi-session, Personalized Cognitive Bias Modification for Thought-Action-Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Han Joo Lee (Other)
Collaborators: Psi Chi (Other)
Responsible Party: Sponsor-Investigator, Han Joo Lee, Professor, University of Wisconsin, Milwaukee
Organization: University of Wisconsin, Milwaukee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWM 24.060
Record Dates: First submitted 2024-11-21; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: OCD
Keywords: Cognitive Bias Modification; Personalization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive Bias Modification for Thought-Action-Fusion (CBM-TAF) (Experimental): CBM-TAF will employ an ambiguous sentence-completion task, where participants have to fill in a missing letter in a fragmented word and resolve emotional ambiguity of a given scenario. At the beginning of each training session, participants will watch a brief animated video about TAF, OCD, and modifying TAF. Each training session will consist of 40 scenarios, which will take about 20 minutes to complete. There will be a total of 6 sessions (2x/week for 3 weeks).
  Interventions: Behavioral: CBM-TAF
- Cognitive Bias Modification for Stress Management Psychoeducation (CBM-SMP) (Active Comparator): Similar to CBM-TAF, CBM-SMP will employ an ambiguous sentence-completion task, where participants have to fill in a missing letter in a fragmented word. However, the content of scenarios in CBM-SMP will focus on general stress management techniques. At the beginning of each training session, participants will watch a brief animated video about OCD and stress management techniques. Each training session will consist of 40 scenarios, which will take about 20 minutes to complete. There will be a total of 6 sessions (2x/week for 3 weeks).
  Interventions: Behavioral: CBM-SMP
- Waitlist (WL) (No Intervention): Participants in WL group will only complete weekly assessment measures without engaging in any training sessions.

INTERVENTIONS:
Behavioral: CBM-TAF — CBM-TAF aims to modify TAF by training participants to adopt an interpretation style that is inconsistent with TAF (i.e., having unwanted thoughts is not morally equivalent to acting upon them and/or having unwanted thoughts does not increase the likelihood of feared events happening in real life). To personalize the training, CBM-TAF is designed to address 4 subtypes of OCD (as defined by Dimensional Obsessive-Compulsive Scale; Abramowitz et al., 2010), each of which targets either TAF-moral or TAF-likelihood. Participants will indicate two OCD subtypes that are most relevant to their experiences and only complete scenarios that correspond to their chosen subtypes. For each scenario, participants are instructed to enter a missing letter in a fragmented word and resolve its emotional ambiguity. After then, participants will answer a True/False question related to the given scenario to verify their comprehension and consolidate their acquisition of healthier interpretation style.
  Arms: Cognitive Bias Modification for Thought-Action-Fusion (CBM-TAF)
Behavioral: CBM-SMP — CBM-SMP is a comparable intervention to CBM-TAF (Siwiec et al., 2023), which aims to provide general education about stress and stress management techniques. It is identical to CBM-TAF in terms of its administration, except for the content of scenarios included in training sessions. For each scenario, participants are instructed to enter a missing letter in a fragmented word. After then, participants will answer a True/False question related to the given scenario in order to verify their comprehension.
  Arms: Cognitive Bias Modification for Stress Management Psychoeducation (CBM-SMP)

SUMMARY:
Thought-Action-Fusion (TAF) is a cognitive bias that posits (1) having unwanted thoughts is morally equivalent to acting upon the thoughts (TAF-Moral; e.g., "Thinking about harming a child is as immoral as actually harming a child") and (2) having unwanted thoughts will increase the likelihood of the thoughts happening in real life (TAF-Likelihood; e.g., "My mother will get into a car accident, because I thought about it"). Given its central role in the development and maintenance of OCD, TAF has emerged as a potential treatment target for obsessive-compulsive disorder (OCD). Previous research has demonstrated that TAF is indeed a malleable construct. This study aims to examine the effects of a multi-session, personalized cognitive bias modification (CBM) for thought-action-fusion (TAF) on improving obsessive-compulsive (OC) symptoms in a college sample.

DETAILED DESCRIPTION:
All participants will be randomized into three groups: 1) CBM-TAF, 2) CBM-SMP (stress management psychoeducation), and 3) WL (waitlist). Participants randomized into either of the training groups (CBM-TAF or CBM-SMP) will complete a total of 6 training sessions (2x/week for 3 weeks), which employ the ambiguous-sentence completion task. To strengthen the training effect, participants will watch brief animated videos about TAF (CBM-TAF) or stress management (CBM-SMP) at the beginning of each session. Participants randomized into the WL group will only complete weekly assessments without any training sessions. All participants will complete pre-, post-training and 1-month follow-up assessments. All training sessions and assessments will be housed on a mobile-based web platform.

ELIGIBILITY:
Inclusion Criteria:

* A score of 18 or higher on the Dimensional Obsessive-Compulsive Scale (DOCS)
* Aged 18 or higher
* Access to a mobile device (i.e., smartphone)

Exclusion Criteria:

* Self-reported visual impairment that cannot be adjusted and will prevent them from clearly recognizing words and pictures on mobile screen
* Self-reported history of a bipolar disorder or psychotic disorder on a Diagnostic History Scale (DHS)
* Inability to adequately understand the study procedure as determined by the responses to comprehension questions provided at the time of the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Thought-Action-Fusion Scale (TAFS) at Pre-, Post-, and 1MFU | Pre-training (before 1st training session), Post-training (at the end of 6th training session, 3 weeks after the 1st training session on average), 1-Month Follow-Up (1 month after the 6th training session)
  The Thought-Action-Fusion Scale (TAFS; Shafran et al., 1996) is a 19-item measure, which assesses the presence and severity of TAF among adults. The measure uses a 5-point Likert scale, which ranges from 0 (Disagree Strongly) to 4 (Agree Strongly) with 12 items assessing TAF-moral, 3 items assessing TAF-likelihood-self, and 4 items assessing TAF-likelihood-others. The measure generates three scores (TAF-total, TAF-Moral, TAF-likelihood) and higher scores indicate higher severity.
Dimensional Obsessive-Compulsive Scale (DOCS) at Pre-, Post-, and 1MFU | Pre-training (before 1st training session), Post-training (at the end of 6th training session, 3 weeks after the 1st training session on average), 1-Month Follow-Up (1 month after the 6th training session)
  Dimensional Obsessive-Compulsive Scale (DOCS; Abramowitz et al., 2010) is a 20-item self-report measure, which assesses the severity of four dimensions of obsessive-compulsive symptoms among adults: 1) Concerns about Germs and Contamination, 2) Concerns about being Responsible for Harm, Injury, or Bad Luck, 3) Unacceptable thoughts (e.g., sex, immorality, violence), and 4) Concerns about Symmetry, Completeness, and the Need for Things to be "Just Right". The measure uses a 4-point Likert Scale, and the total score of DOCS ranges from 0 to 80. A cutoff score of 21 was established to distinguish individuals with clinically severe OC symptoms by the measure developers (Abramowitz et al., 2010).

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS-21) at Pre-, Post-, and 1MFU | Pre-training (before 1st training session), Post-training (at the end of 6th training session, 3 weeks after the 1st training session on average), 1-Month Follow-Up (1 month after the 6th training session)
  Depression, Anxiety, and Stress Scale (DASS-21; Lovibond & Lovibond, 1995) is a 21-item self-report measure, which assesses symptoms of depression, anxiety, and stress. The measure uses a 4-point Likert scale, which ranges from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). Higher scores indicate more severe depression, anxiety, and stress symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hanjoo Lee, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- UWM Anxiety Disorders Laboratory, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathews A, Mackintosh B. Induced emotional interpretation bias and anxiety. J Abnorm Psychol. 2000 Nov;109(4):602-15. PMID 11195984
- [Background] Abramowitz JS, Deacon BJ, Olatunji BO, Wheaton MG, Berman NC, Losardo D, Timpano KR, McGrath PB, Riemann BC, Adams T, Bjorgvinsson T, Storch EA, Hale LR. Assessment of obsessive-compulsive symptom dimensions: development and evaluation of the Dimensional Obsessive-Compulsive Scale. Psychol Assess. 2010 Mar;22(1):180-98. doi: 10.1037/a0018260. PMID 20230164
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Shafran R, Thordarson DS, Rachman S. Thought-action fusion in obsessive compulsive disorder. Journal of Anxiety Disorders. 1996; 10(5), 379-391.
- [Background] Siwiec S, Bodhy S, Lotfi S, Lee, HJ. Cognitive bias modification for thought-action fusion: A placebo-controlled randomized experimental trial. Journal of Obsessive-Compulsive and Related Disorders. 2023; 37, 100787.